CLINICAL TRIAL: NCT00033592
Title: Phase III Trial Comparing Nicotine Inhaler Versus Bupropion Versus Nicotine Inhaler Plus Bupropion For Smoking Cessation Efficacy And Relapse Prevention
Brief Title: Comparison of Nicotine Inhaler and/or Bupropion in Helping People to Stop Smoking and Prevent the Recurrence of Smoking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NCCTG-N99C4; CDR0000069303 (Registry Identifier: PDQ (Physician Data Query)); NCI-P02-0220
Record Dates: First submitted 2002-04-09; First posted 2004-02-06 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Bupropion; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (15):
- Arm I: nicotine inhaler cartridges (Experimental): Participants receive 6-16 nicotine inhaler cartridges per day. Treatment continues for 12 weeks. After 12 weeks, participants are randomized a second time based on whether they continue to smoke or are smoke-free.
  Participants randomized to arm I who continue to smoke are randomized to one of two treatment arms Arm IV or Arm V. Participants randomized to arm I who are smoke-free are randomized to one of two treatment arms Arm VIII or Arm IX.
  Interventions: Drug: nicotine
- Arm II: bupropion (Experimental): Participants receive oral bupropion 1-2 times daily.
  Treatment continues for 12 weeks. After 12 weeks, participants are randomized a second time based on whether they continue to smoke or are smoke-free. After 12 weeks, participants are randomized a second time based on whether they continue to smoke or are smoke-free.
  Participants randomized to arm II who continue to smoke are randomized to one of two treatment arms Arm VI or Arm VII. Participants randomized to arm II who are smoke-free are randomized to one of two treatment arms Arm Arm X or Arm XI.
  Interventions: Drug: bupropion hydrochloride
- Arm III: nicotine inhaler cartridges (Experimental): Participants receive 6-16 nicotine inhaler cartridges per day and oral bupropion 1-2 times daily. Treatment continues for 12 weeks. After 12 weeks, participants are randomized a second time based on whether they continue to smoke or are smoke-free.
  Participants randomized to arm III who continue to smoke do not receive any further therapy. Participants randomized to arm III who are smoke-free are randomized to one of four treatment arms Arm XII, Arm XIII, Arm XIV or Arm XV.
  Interventions: Drug: nicotine
- Arm IV: bupropion (Experimental): Participants receive oral bupropion 1-2 times daily for 12 weeks.
  All participants are followed every month for 6 months.
  Interventions: Drug: bupropion hydrochloride
- Arm V: placebo (Placebo Comparator): Participants receive oral placebo 1-2 times daily for 12 weeks.
  All participants are followed every month for 6 months.
  Interventions: Other: placebo
- Arm VI: nicotine inhaler cartridges (Experimental): Participants receive 6-16 nicotine inhaler cartridges per day for 12 weeks.
  All participants are followed every month for 6 months.
  Interventions: Drug: nicotine
- Arm VII: placebo inhaler (Placebo Comparator): Participants receive 6-16 placebo inhaler cartridges per day for 12 weeks.
  All participants are followed every month for 6 months.
  Interventions: Other: placebo
- Arm VIII: nicotine inhaler cartridges (Experimental): Participants receive 6-16 nicotine inhaler cartridges per day for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Drug: nicotine
- Arm IX: placebo inhaler cartridges (Placebo Comparator): Participants receive 6-16 placebo inhaler cartridges per day for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Other: placebo
- Arm X: bupropion (Experimental): Participants receive oral bupropion 1-2 times daily for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Drug: bupropion hydrochloride
- Arm XI: placebo (Placebo Comparator): Participants receive oral placebo 1-2 times daily for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Other: placebo
- Arm XII: nicotine inhaler cartridges (Experimental): Participants receive 6-16 nicotine inhaler cartridges per day and oral placebo 1-2 times daily for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Drug: nicotine
- Arm XIII: placebo inhaler cartridges (Placebo Comparator): Participants receive 6-16 placebo inhaler cartridges per day and oral bupropion 1-2 times daily for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Other: placebo
- Arm XIV: nicotine inhaler cartridges (Experimental): Participants receive 6-16 nicotine inhaler cartridges per day and oral bupropion 1-2 times daily for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Drug: nicotine
- Arm XV: placebo inhaler cartridges (Placebo Comparator): Participants receive 6-16 placebo inhaler cartridges per day and oral placebo 1-2 times daily for 40 weeks.
  All participants are followed every month for 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo
  Arms: Arm IX: placebo inhaler cartridges; Arm V: placebo; Arm VII: placebo inhaler; Arm XI: placebo; Arm XIII: placebo inhaler cartridges; Arm XV: placebo inhaler cartridges
Drug: bupropion hydrochloride
  Arms: Arm II: bupropion; Arm IV: bupropion; Arm X: bupropion
Drug: nicotine
  Arms: Arm I: nicotine inhaler cartridges; Arm III: nicotine inhaler cartridges; Arm VI: nicotine inhaler cartridges; Arm VIII: nicotine inhaler cartridges; Arm XII: nicotine inhaler cartridges; Arm XIV: nicotine inhaler cartridges

SUMMARY:
RATIONALE: Use of a nicotine inhaler and/or bupropion may be effective in helping people stop smoking and prevent them from starting smoking again. It is not yet known whether a nicotine inhaler or bupropion are more effective alone or combined for stopping smoking.

PURPOSE: Randomized phase III trial to compare the effectiveness of the nicotine inhaler or bupropion alone to that of the nicotine inhaler combined with bupropion in helping people to stop smoking and prevent starting smoking again.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effectiveness of nicotine inhaler vs bupropion vs nicotine inhaler plus bupropion on smoking cessation and prevention of relapse in participants who currently smoke. II. Compare the reduction in the rate of relapse to smoking after initial abstinence in participants treated long term with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to gender, cigarettes smoked per day at time of screening (10-39 vs 40 or more), and total length of smoking in years (less than 5 vs 5-9 vs 10 or more). Participants are randomized to one of three treatment arms. Arm I: Participants receive 6-16 nicotine inhaler cartridges per day. Arm II: Participants receive oral bupropion 1-2 times daily. Arm III: Participants receive 6-16 nicotine inhaler cartridges per day and oral bupropion 1-2 times daily. In all arms, treatment continues for 12 weeks. After 12 weeks, participants are randomized a second time based on whether they continue to smoke or are smoke-free. Participants randomized to arm I who continue to smoke are randomized to one of two treatment arms. Arm IV: Participants receive oral bupropion 1-2 times daily for 12 weeks Arm V: Participants receive oral placebo 1-2 times daily for 12 weeks. Participants randomized to arm II who continue to smoke are randomized to one of two treatment arms. Arm VI: Participants receive 6-16 nicotine inhaler cartridges per day for 12 weeks. Arm VII: Participants receive 6-16 placebo inhaler cartridges per day for 12 weeks. Participants randomized to arm III who continue to smoke do not receive any further therapy. Participants randomized to arm I who are smoke-free are randomized to one of two treatment arms. Arm VIII: Participants receive 6-16 nicotine inhaler cartridges per day for 40 weeks. Arm IX: Participants receive 6-16 placebo inhaler cartridges per day for 40 weeks. Participants randomized to arm II who are smoke-free are randomized to one of two treatment arms. Arm X: Participants receive oral bupropion 1-2 times daily for 40 weeks. Arm XI: Participants receive oral placebo 1-2 times daily for 40 weeks. Participants randomized to arm III who are smoke-free are randomized to one of four treatment arms. Arm XII: Participants receive 6-16 nicotine inhaler cartridges per day and oral placebo 1-2 times daily for 40 weeks. Arm XIII: Participants receive 6-16 placebo inhaler cartridges per day and oral bupropion 1-2 times daily for 40 weeks. Arm XIV: Participants receive 6-16 nicotine inhaler cartridges per day and oral bupropion 1-2 times daily for 40 weeks. Arm XV: Participants receive 6-16 placebo inhaler cartridges per day and oral placebo 1-2 times daily for 40 weeks. All participants are followed every month for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Currently smoking at least 10 cigarettes per day Smoked regularly for the past year Motivated to use study medication More than 30 days since prior use of tobacco products other than cigarettes (e.g., smokeless tobacco, pipes, cigars, or snuff) No active chemical dependence of drug other than nicotine (e.g., alcohol, marijuana, cocaine, heroin, or other illicit drugs) within the past year

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No unstable angina, myocardial infarction, or cardiac arrhythmias within the past 3 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for at least 3 months prior to and during study Good health by medical history No history of seizure disorder No epilepsy No prior serious head trauma or other predisposing factors to seizures (e.g., alcohol withdrawal, febrile seizures during childhood, brain tumor, cerebrovascular accident, or family history of idiopathic seizure disorder) No known hypersensitivity or allergy to nicotine, menthol, or bupropion No prior or concurrent diagnosis of bulimia or anorexia nervosa No other member of household currently enrolled on this study No bipolar disorder, psychosis, or schizophrenia

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: More than 30 days since prior systemic steroids Radiotherapy: Not specified Surgery: Not specified Other: More than 30 days since other prior behavioral or pharmacologic smoking- cessation program (e.g., behavioral therapy, nicotine replacement therapy, clonidine, bupropion, nortriptyline, or doxepin) More than 30 days since prior investigational drugs More than 30 days since prior antipsychotics or antidepressants More than 30 days since prior theophylline More than 30 days since prior monoamine oxidase inhibitor More than 30 days since prior medication containing bupropion No concurrent antiepileptic medications No concurrent medications known to lower seizure threshold No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1708 (Actual)
Dates: Start 2002-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Prevention in relapse | Up to 6 months

SECONDARY OUTCOMES:
Reduction in the rate of relapse | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Hurt, MD, Study Chair — Mayo Clinic
Locations (25):
- United States (24):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961